CLINICAL TRIAL: NCT06515444
Title: 10-minutes Project: Experimental Evaluation of the 10-minute Program to Foster Socioemotional Competence of Children in Third Grade and Their Teachers
Brief Title: Experimental Evaluation of a Program to Foster Socioemotional Competence of Children in Third Grade and Their Teachers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de los Andes, Chile (Other)
Collaborators: Agencia Nacional de Investigación y Desarrollo (Other)
Responsible Party: Principal Investigator, Barbara Hanisch Cerda, PhD, Universidad de los Andes, Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEC2024029
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Social Skills; Emotion Regulation
MeSH Terms: conditions — Social Skills; Emotional Regulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 10 minutes only (Experimental): Group will only receive a socioemotional development material for teachers to implement with their students
  Interventions: Behavioral: 10 minutes program
- 10 minutes plus (Experimental): Group will receive socioemotioanl devleopment material for teachers to implement with their students plus professional development for teachers
  Interventions: Behavioral: 10 minutes program; Behavioral: 1 hour PD program
- Delayed (Other): While intervention in arms 1 and 2, this arm will not receive internvention. It will receive the 10 minutes plus, once the other two arms have their second year follow up measure.
  Interventions: Behavioral: 10 minutes program; Behavioral: 1 hour PD program

INTERVENTIONS:
Behavioral: 10 minutes program — The curriculum component offers 10-minute daily doses of activities targeting the development of eight socioemotional competences in children: (i) emotional knowledge and management, (ii) developing a healthy identity, (iii) establishing and maintaining positive relationships, (iv) feeling and showing empathy, (v) establishing and reaching goals, (vi) responsible decision-making, (vii) contributing to the community and (viii) developing spirituality. The activities do not require the teacher to plan or to prepare material for the students.
Behavioral: 1 hour PD program — The professional development (PD) component is a 1-hour dose of activities targeting each of the eight SECs on which the curriculum focuses. The focus of PD is not to teach about SEC development in children but to develop SEC in teachers. Thus, this is an 8-hour PD program distributed throughout the academic year.
  Arms: 10 minutes plus; Delayed

SUMMARY:
The 10-minutes project is an experimental study to assess the impact of a SEL program for children in 3th and 4th grade and their teachers called 10-minutes.

The program is a curriculum that provides 10-minute activities (thus the name) for children to be implemented by the teachers daily throughout the school year. The activities do not require prior knowledge of teachers on SEL development, nor planning or material preparation.

The 10-minute project is a quantitative study developed to evaluate whether the 10-minute curriculum and an expanded version with professional development activities for teachers or counselors, 10-minute plus, at third grade would improve students and teachers' socioemotional competence. The randomized control trail involves 30 schools in Chile, matched on socioeconomic measures, size, and urban/rural conditions, assigned randomly to 1 of 3 conditions. Ten schools will receive 10-minutes only, the SEL curriculum taught by teachers or school counselors, during the 2024 and 2025 school years. Ten schools will receive 10-minutes plus during the 2024 school year. Ten schools will serve as "delayed program" control, which will have the opportunity to receive the program (10-minutes plus) after the final follow-up. To examine the possibility of fade-out of the effects of the SEL intervention on students, the first experimental condition (10-minutes only) will be randomly divided into two groups, one will receive the intervention for one year only, whereas the second one will receive the intervention for two consecutive years.

It is expected the program will yield positive effects on the experimental groups (both students and teachers), and effects are expected to be greater in the group offered the 10-minutes plus intervention which entails both a curriculum for children and professional development for teachers, than the effects in the group offered the 10-minutes curriculum exclusively. If the program proves to be effective, then cost-benefit analyses will follow to assess the efficiency of the program. The estimated benefits of the program are expected to be lower than the costs.

DETAILED DESCRIPTION:
Over the last 20 years the science of learning and economics of education has uplifted the relevance of socioemotional competence both for learning and other societal outcomes. Findings from neurobiology have illuminated how environmental factors such as poverty, exposure to stress or experiencing trauma, affect children's development of brain systems that support neurocognitive functions such as language, memory and self-regulation and therefore affecting their behavior, lifelong learning, and health (Immordino-Yang & Damasio, 2007; Twardosz & Lutzker, 2010; Noble, 2014; Chapko, 2015; Kolb & Gibb, 2015; Thomason & Marusak, 2017). Findings from the economics of education consistently indicates positive relationships between noncognitive skills and societal outcomes such as educational attainment (Farrington et al., 2012; Levin, 2012; Garcia, 2015), labor productivity and adult earnings (Casner-Lotto & Barrington, 2006; Heckman, Stixrud & Urzua, 2006; Murnane et al., 2001), and civic participation (Almlund, Duckworth, Heckman & Kautz, 2011). This has led educators to pursue new strategies to support the social and emotional competence of children as well as their academic learning. Socioemotional learning (SEL hereafter) is the process through which individuals acquire socioemotional competence, the "process through which all young people and adults acquire and apply the knowledge, skills, and attitudes to develop healthy identities, manage emotions and achieve personal and collective goals, feel and show empathy for others, establish and maintain supportive relationships, and make responsible and caring decisions" (Niemi, 2020).

The 10-minutes project is a pilot study to assess the impact of a SEL program for children in 3th and 4th grade and their teachers called 10-minutes.

The program is a curriculum that provides 10-minute activities (thus the name) for children to be implemented by the teachers daily throughout the school year. The activities do not require prior knowledge of teachers on SEL development, nor planning or material preparation. Each activity is presented along with knowledge for teachers on how to develop socioemotional skills in children. The curriculum is complemented by professional development for teachers on the development of their own socioemotional competencies.

The 10-minute project is a pilot study, primarily exploratory. It will provide data on the feasibility of the program, and its acceptability. The 10-minute project also has a quantitative study developed to evaluate whether the 10-minute curriculum and an expanded version with professional development activities for teachers or counselors, 10-minute plus, at third grade would improve students and teachers' socioemotional competence. The randomized control trail involves 30 schools in Chile, matched on socioeconomic measures, size, and urban/rural conditions, assigned randomly to 1 of 3 conditions. Ten schools will receive 10-minutes only, the SEL curriculum taught by teachers or school counselors, during the 2024 and 2025 school years. Ten schools will receive 10-minutes plus during the 2024 school year. Ten schools will serve as "delayed program" control, which will have the opportunity to receive the program (10-minutes plus) after the final follow-up. To examine the possibility of fade-out of the effects of the SEL intervention on students, the first experimental condition (10-minutes only) will be randomly divided into two groups, one will receive the intervention for one year only, whereas the second one will receive the intervention for two consecutive years. Surveys will be used to collect data on student, classroom, and teacher outcomes in the 30 schools in fall 2024 (baseline), spring 2024 (first follow-up), and among fourth grade students in the same schools in spring 2025 (final follow-up). The intervention will take place after the baseline data is collected in March and April 2024.

It is expected the program will yield positive effects on the experimental groups (both students and teachers), and effects are expected to be greater in the group offered the 10-minutes plus intervention which entails both a curriculum for children and professional development for teachers, than the effects in the group offered the 10-minutes curriculum exclusively. If the program proves to be effective, then cost-benefit analyses will follow to assess the efficiency of the program. The estimated benefits of the program are expected to be lower than the costs.

Why this program and study matters? This program and study are relevant for two main reasons: First, children and adults are facing a mental health crisis in Chile and elsewhere (Humphreys & Irarrazaval, 2022; World Health Organization, 2022), and SEL programs have proven to be an effective way to increase children and adults' socioemotional competence (Durlak et al., in press), fundamental skills to cope with environmental stressors and daily challenges. Second, Chilean teachers have received little to no training in pre-service education (Milici & Alcalay, 2020) and admit not having the necessary tools to tackle SEL in schools (Berger et al., 2009). This project presents an intervention that helps tackle both challenges and present a robust study design to argue for the causal impact of the intervention on children's and teachers' socioemotional competencies.

ELIGIBILITY:
Inclusion Criteria:

* . The inclusion criteria for schools: at least one third and one fourth grade class.

Exclusion Criteria:

* The exclusion criteria for schools are as follows: schools implementing a similar intervention in grades 3 and 4, and special needs schools.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2024-07-22 (Estimated); Primary Completion 2026-12-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Learning characteristics, leadership, motivation, communication, and planning skills. | Months 1, 5 and 12
  The Scales for Rating the Behavioral Characteristics of Superior Students developed by Renzulli et al. (2002) will be used. This scale has 14 subscales. Only 5 will be used: leadership, learning characteristics, motivation, communication, and planning skills. The other scales refer to learning behavior in specific disciplines (such as arts, music, science, etc.) and that is why they will not be used. The items of these scales will be responded by parents.
Self-control | Months 1, 5 and 12
  will be assessed using the Impulsivity Scale for Children (ISC). This is an 8-item survey responded by children that assesses the inability to regulate behavior, attention, and emotions in specific goals (Tsukayama, Duckworth & Kim, 2013).
Grit | Months 1, 5 and 12
  The 10-item likert scale that measures perseverance, the Oviedo Grit Scale (OGS; Postigo, Cuesta, García-Cueto et al., 2021) will be used. The scale has been adapted to Chile (reliability = 0.92; Postigo, Barria, Cuesta, Garcia-Cueto, 2023).
Mindset | Months 1, 5 and 12
  Whether children view intelligence as a fixed trait rather than a trait that can be improved will be assessed using a 3-item scale developed by Dweck, Chiu and Hong (1995), widely used in Chile with an internal consistency of 0.86 (Claro, Paunesku & Dweck, 2016).
Pro-social attitude | Months 1, 5 and 12
  will be assessed using the 18-item Empathy Questionnaire for Children and Adolescents (EmQue-CA) developed by Overgaauw, and colleagues (2017).
Behavioral difficulties | Months 1, 5 and 12
  will be assessed using the 20-item parental or teacher survey Strengths and Difficulties Questionnaire (SDQ) developed by Goodman (1997). The version for children was validated in Chile by Gaete et al. (2018) with internal consistency fluctuating between .76 and .85.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Hanisch-Cerda, PhD, Principal Investigator — Universidad de los Andes, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hanisch-Cerda B, Benitez-Yavar D. Enhancing socioemotional competencies: protocol for a three-arm cluster randomized controlled trial of a daily program for third graders and educators. Trials. 2025 Dec 24;26(1):580. doi: 10.1186/s13063-025-09183-0. PMID 41444899